CLINICAL TRIAL: NCT05589558
Title: Prospective Comparison of the Four Biopsy Methods for Prostate Cancer Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Professor, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sechenov-four_biopsies
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: prostate cancer; fusion biopsy; cognitive biopsy; transrectal ultrasound biopsy; transperineal template mapping biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gene Fusion

STUDY DESIGN:
Intervention Model Description: First step: the "unblinded" urologist №1 performed a fusion and transpeineal template mapping biopsy. Second step: the "blinded" urologist №2 performed TRUS-guided and cognitive biopsy. All specimens were obtained within a single procedure.
Masking Description: The "blinded" urologist performed TRUS-guided and cognitive biopsy without prior knowledge about MRI results
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with suspected prostate cancer underwent 4 biopsy methods (Experimental): Patients with suspected prostate cancer consequently underwent TRUS-guided, cognitive, fusion and transperineal template mapping biopsy
  Interventions: Procedure: consequently performed 4 biopsy methods (TRUS-guided biopsy, cognitive, fusion and transperineal template mapping biopsy)

INTERVENTIONS:
Procedure: consequently performed 4 biopsy methods (TRUS-guided biopsy, cognitive, fusion and transperineal template mapping biopsy) — TRUS-guided biopsy - extensive number of biopsies taken transrectally involving peripheral and transitional zones (8-12 cores); cognitive biopsy - targeted biopsy with MRI information and TRUS guidance but without fusion technology (2-4 cores); fusion biopsy - targeted biopsy with MRI information using MRI/TRUS fusion technology (2-4 core); transperineal template mapping biopsy - systematic transperineal TRUS-guided biopsy with special template use to aid accurate placement of biopsy needles (more than 20 cores).

SUMMARY:
The aim of this study is to compare clinically significant prostate cancer detection rate by the 4 biopsy methods: TRUS-guided, cognitive, fusion and transperineal template mapping biopsy.

It is recommended to combine MRI-guided biopsy with systematic (TRUS-guided or transperineal template mapping biopsy) biopsy for high yield of prostate cancer diagnosis. Nevertheless, it remains unclear which biopsy combination is more precise for prostate cancer detection.

DETAILED DESCRIPTION:
Taking into consideration the variety of prostate biopsy methods (TRUS-guided, cognitive, fusion and transperineal template mapping biopsy), the issue of indications for each of them remains unresolved. Current EAU guidelines recommend combining MRI-guided biopsy with systematic (TRUS-guided or transperineal template mapping biopsy) one for high yield of prostate cancer diagnosis. Nevertheless, it also remains unclear which biopsy combination is more precise for prostate cancer detection.

This is a prospective single-arm study.

All patients underwent prostate TRUS examination and mpMRI. Suspicious lesion found on MRI were classified with the Pi-RADS v2.1. First step: the "unblinded" urologist №1 performed a fusion and transperineal template mapping biopsy. Second step: the "blinded" urologist №2 performed TRUS-guided and cognitive biopsy.

Objectives of the study: to determine clinically significant prostate cancer detection rate, overall cancer detection rate, clinically insignificant prostate cancer detection rate, sampling efficiency (positive biopsy cores' number, maximum cancer core length (MCCL)). Results were calculated for each biopsy method separately and for combinations of TRUS-guided and cognitive biopsy (combination №1) and fusion and transperineal template mapping biopsy (combination №2).

ELIGIBILITY:
Inclusion Criteria:

* PSA >2 ng/mL, and/or positive digital rectal examination (DRE), and/or suspicious lesion on TRUS
* Pi-RADSv2.1 ≥3 score

Exclusion Criteria:

* previously diagnosed PCa;
* acute prostatitis within the last 3 months;
* 5-α reductase inhibitors therapy within the last 6 months;
* extracapsular extension;
* prostate volume ≥80 cc;
* contraindications for mpMRI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Clinically significant prostate cancer detection rate | 2 weeks after performed 4 biopsy methods
  Ratio of patients with preoperative Pi-RADS ≥3 with defined clinically significant prostate cancer (ISUP ≥2) in relation to total number of patients

SECONDARY OUTCOMES:
Overall prostate cancer detection rate | 2 weeks after performed 4 biopsy methods
  Ratio of patients with preoperative Pi-RADS ≥3 with defined prostate cancer in relation to total number of patients
Clinically insignificant prostate cancer detection rate | 2 weeks after performed 4 biopsy methods
  Ratio of patients with preoperative Pi-RADS ≥3 with defined clinically insignificant prostate cancer (ISUP 1) in relation to total number of patients
Positive biopsy cores' number | 2 weeks after performed 4 biopsy methods
  Ratio of cores with detected prostate cancer in relation to overall numbers of cores
Maximum cancer core length | 2 weeks after performed 4 biopsy methods
  Median length of core with prostate cancer in realtion to whole biopsy core
Number of missed clinically significant prostate cancer | 2 weeks after performed 4 biopsy methods
  Ratio of patients with preoperative Pi-RADS ≥3 with downgraded ISUP score in relation to maximum ISUP score obtained among biopsies
Added value of prostate cancer | 2 weeks after performed 4 biopsy methods
  Ratio of patients with preoperative Pi-RADS ≥3 with upgraded ISUP score in relation to maximum ISUP score obtained among biopsies
Predicting factors of PCa detection | 2 weeks after performed 4 biopsy methods
  Prognostic factors of clinically significant and overall prostate cancer detection rate
Comparison of biopsies and post-prostatectomy pathological results | 2 weeks after radical prostatectomy
  Gleason score obtained within biopsy and the post-prostatectomy pathology

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

REFERENCES:
- [Background] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724